CLINICAL TRIAL: NCT07202819
Title: Does Neoadjuvant Chemotherapy Affect the Accuracy of Magnetic Resonance Imaging Before Radical Cystectomy? A Randomized Controlled Trial.
Brief Title: Effect of Neoadjuvant Chemotherapy on MRI Accuracy Before Cystectomy
Acronym: "NAC-MRI"
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amr Esam Saad Mohamed Darwish, Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PreIRB-Assiut-URO001
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Muscle Invasive Bladder Cancer
MeSH Terms: interventions — Neoadjuvant Therapy; Cystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neoadjuvant Chemotherapy Arm (Active Comparator): Participants in this arm will receive standard-of-care neoadjuvant chemotherapy (NAC) before undergoing radical cystectomy for muscle-invasive bladder cancer (MIBC). MRI will be performed post-NAC for local tumor restaging, and the results will be compared to histopathology to evaluate the diagnostic accuracy of MRI.
  Interventions: Drug: Neoadjuvant Chemotherapy; Procedure: Radical Cystectomy
- Radical cystectomy-Only arm (Active Comparator): Participants in this arm will undergo immediate radical cystectomy without receiving neoadjuvant chemotherapy. MRI will be performed preoperatively for local tumor staging, and results will be compared with post-surgical histopathology to assess the accuracy of MRI in this setting.
  Interventions: Procedure: Radical Cystectomy

INTERVENTIONS:
Drug: Neoadjuvant Chemotherapy — Standard neoadjuvant chemotherapy for muscle-invasive bladder cancer, typically consisting of cisplatin-based regimens such as MVAC (methotrexate, vinblastine, doxorubicin, and cisplatin) or gemcitabine and cisplatin. Administered prior to radical cystectomy to shrink the tumor and improve surgical outcomes. The post-treatment MRI findings will be analyzed for correlation with histopathological results after surgery.
  Other Names: NAC
  Arms: Neoadjuvant Chemotherapy Arm
Procedure: Radical Cystectomy — Surgical removal of the urinary bladder, typically performed in patients with muscle-invasive bladder cancer. In this study, participants in both arms will undergo radical cystectomy, either directly or following neoadjuvant chemotherapy. Histopathological examination of surgical specimens will be compared with MRI findings for staging accuracy assessment.
  Other Names: RC

SUMMARY:
The goal of this clinical trial is to learn if neoadjuvant chemotherapy (NAC) affects the accuracy of magnetic resonance imaging (MRI) in staging muscle-invasive bladder cancer (MIBC). This study will also assess how tissue changes induced by NAC impact MRI interpretation. The main questions it aims to answer are:

Does NAC compromise the accuracy of MRI in staging MIBC?

Does NAC-induced tissue change affect the reliability of MRI in tumor assessment?

Researchers will compare MRI staging accuracy in MIBC patients who received NAC to those who went directly to surgery, to see if NAC impacts MRI's diagnostic performance.

Participants will:

Undergo MRI scanning before surgery

Receive either NAC or go directly to surgery, depending on their group assignment

Have their MRI results compared to histopathological outcomes after surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cT2 urothelial carcinoma of the urinary bladder, according to the TNM classification, who give informed, written consent on participation in the study and approve all its requirements.

Exclusion Criteria:

* Patients who have received pelvic radiotherapy.
* Previous open or laparoscopic pelvic surgery.
* Patients with contraindications to MRI.
* Patients who are unfit for or refuse radical cystectomy.
* Ineligibility to cisplatin.
* squamous differentiation in the histopathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Compare the accuracy of MRI between patients who received and those who didn't receive NAC | At the time of radical cystectomy and final histopathology report (approximately 3 to 6 months after starting NAC)
  This outcome aims to evaluate and compare the diagnostic accuracy of MRI in detecting tumor stage in bladder cancer patients who underwent NAC prior to radical cystectomy versus those who did not receive NAC.

CONTACTS AND LOCATIONS:
Overall Officials: Amr Darwish, Lecturer, Principal Investigator — Assiut University
Locations (1):
- Urology Department, Faculty of Medicine, Assiut University, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No